CLINICAL TRIAL: NCT01993212
Title: A Randomized, Double Blind, Placebo-Controlled, Multi-Center Phase III Study in Men With Acquired Hypogonadotropic Hypogonadism to Compare Changes in Testosterone and Sperm Concentration Following Treatment With 12.5 mg or 25 mg Androxal or AndroGel 1.62%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZA-304
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Secondary Hypogonadism
Keywords: Low Testosterone
MeSH Terms: conditions — Hypogonadism | interventions — Enclomiphene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Androxal Placebo and Gel Placebo
  Interventions: Drug: Placebo Capsules; Drug: Placebo Gel
- AndroGel Treatment (Active Comparator): AndroGel 1.62% and Placebo Capsules
  Interventions: Drug: AndroGel 1.62%; Drug: Placebo Capsules
- Androxal Treatment (Experimental): Androxal 12.5 mg or 25mg and Placebo Gel
  Interventions: Drug: Androxal 12.5 mg or 25 mg; Drug: Placebo Gel

INTERVENTIONS:
Drug: Androxal 12.5 mg or 25 mg
  Arms: Androxal Treatment
Drug: AndroGel 1.62%
  Arms: AndroGel Treatment
Drug: Placebo Capsules
  Arms: AndroGel Treatment; Placebo
Drug: Placebo Gel
  Arms: Androxal Treatment; Placebo

SUMMARY:
This is a Randomized, Double Blind, Placebo-Controlled, Multi-Center Phase III Study in Men with Acquired Hypogonadotropic Hypogonadism to Compare Changes in Testosterone and Sperm Concentration Following Treatment with the 12.5 mg or 25 mg Androxal or AndroGel 1.62%.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (BMI 25 to 42 kg/m2 inclusive) males age 18 to 60 inclusive
* Previously or concurrently diagnosed as having secondary hypogonadism characterized as having at least 2 consecutive morning testosterone assessments < 300ng/dL, one of which must be confirmed at Baseline.
* LH < 9.4 mIU/mL (at Visit 1 only)
* Sperm concentration ≥ 15 million per milliliter (assessed at V2 and Baseline). V2 and Baseline measurements must be at least 48 hours apart.
* Ability to complete the study in compliance with the protocol
* Ability to understand and provide written informed consent
* Agreement to provide a total of at least 4 semen samples in a sponsor-approved clinic on 4 separate occasions.

Exclusion Criteria:

* Any prior use of testosterone treatments (injectable, pelleted, transdermal or sublingual) within the last 6 months
* Use of spironolactone, cimetidine, Clomid, 5α-reductase inhibitors, hCG, androgen, estrogen, anabolic steroid, DHEA, or herbal hormone products during the study
* Use of Clomid in the past year
* Any clinically significant laboratory abnormality that does not have prior written sponsor approval. If the sponsor approves subject enrollment, this will not be considered to be a protocol deviation.
* Uncontrolled hypertension or diabetes mellitus based on the Investigator's assessment at baseline. Subjects treated for Type II diabetes will be allowed into the study, if considered clinically stable by the investigator. Newly diagnosed diabetics need to be treated for at least 48 hours before being enrolled in the study.
* A hematocrit >54
* Use of an investigational drug or product, or participation in a drug or medical device research study within 30 days prior to receiving study medication.
* Known hypersensitivity to Clomid
* Symptomatic cataracts (nuclear sclerosis cataract or cortical cataract grade > 2 based on 0-4 scale or any evidence of posterior subcapsular cataract)
* Abnormal fundoscopy exam such as central retinal vein occlusion
* Any condition which in the opinion of the investigator would interfere with the participant's ability to provide informed consent, comply with study instructions, possibly confound interpretation of study results, or endanger the participant if he took part in the study
* Have received a diagnosis of irreversible infertility or compromised fertility (cryptorchism, Kallman Syndrome, primary hypogonadism, vasectomy, or tumors of the pituitary), or history of evaluation or treatment for low fertility
* Current or history of breast cancer
* Current or history of prostate cancer or a suspicion of prostate disease unless ruled out by prostate biopsy, or a PSA>3.6
* Presence or history of known hyperprolactinemia with or without a tumor (prolactin > 20 ng/mL).
* Chronic use of medications such as glucocorticoids (chronic use of inhaled or topical glucocorticoids is acceptable)
* History of drug abuse or chronic narcotic use including methadone
* A recent history of alcoholism or illegal substance or steroid abuse (<2 years) or presence of moderate alcohol use (>21 drinks per week)
* Subjects with known history of HIV and/or Hepatitis C
* Subjects with end stage renal disease
* History of liver disease (including malignancy) or a confirmed AST or ALT >3 times the upper limit of normal
* History of clinically relevant myocardial infarction (within the previous year), unstable angina, symptomatic heart failure, ventricular dysrhythmia or know history of QTc interval prolongation
* History of clinically relevant cerebrovascular disease
* History of venous thromboembolic disease (e.g. deep vein thrombosis or pulmonary embolism)
* History of erythrocytosis or polycythemia
* Subjects unable to provide a semen sample in a sponsor-approved clinic
* Enrollment in a previous Androxal study
* Subjects who have Type I Diabetes

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the proportion of subjects meeting the composite endpoint for normal morning testosterone and semen concentration. | 16 weeks of treatment
  Comparison of the proportion of subjects whose morning testosterone levels are within the normal range [300-1,040 ng/dL] and whose sperm concentration is 15 million/mL or greater following 16 weeks of treatment with Androxal, placebo or AndroGel 1.62%.

SECONDARY OUTCOMES:
Proportion of subjects with mean sperm concentration less than 15 million/mL after 16 weeks of treatment comparing Androxal to placebo in a non-inferiority assessment | 16 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Jacksonville, Florida
  - Albany, New York
  - Raleigh, North Carolina
  - Cleveland, Ohio
  - Medford, Oregon
  - Warwick, Rhode Island
  - Houston, Texas
  - Webster, Texas